CLINICAL TRIAL: NCT06908993
Title: A Randomized Controlled Trial of Tepotinib vs Standard Treatment in Patients With Advanced MET Exon 14 Mutated Non-Small Cell Lung Cancer
Brief Title: Tepotinib vs Standard Treatment in Patients With Advanced MET Exon 14 Mutated Non-Small Cell Lung Cancer Previously Treated
Acronym: COMET
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Intergroupe Francophone de Cancerologie Thoracique (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IFCT-2404; 2024-519971-25-00 (EU CTIS Number)
Record Dates: First submitted 2025-03-27; First posted 2025-04-03 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Advanced Non Small Cell Lung Cancer; MET Exon 14 Mutation
Keywords: Tepotinib; MET Exon 14 Mutation; Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — tepotinib; Pemetrexed; Vinorelbine; Gemcitabine; Docetaxel; Paclitaxel; pembrolizumab; Nivolumab; atezolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Investigator choice treatment (Active Comparator): Investigator's choice treatment among:
  * Monochemotherapy (including pemetrexed, docetaxel, paclitaxel with or without bevacizumab, gemcitabine, vinorelbine),
  * Anti-PD(L)1 agent (including pembrolizumab, nivolumab or atezolizumab),
  * Best supportive care - available only for patients with i) ECOG PS 3 or ii) contraindication to propose a systemic treatment based on an oncogeriatric assessment or confirmed by the local multidisciplinary tumor board.
  The treatment chosen cannot be a treatment already received.
  Interventions: Drug: Pemetrexed (Alimta); Drug: Vinorelbine; Drug: Gemcitabine alone; Drug: Docetaxel; Drug: Paclitaxel; Drug: Pembrolizumab; Drug: Nivolumab; Drug: Atezolizumab
- Tepotinib (Experimental)
  Interventions: Drug: Tepotinib

INTERVENTIONS:
Drug: Tepotinib — Tepotinib will be given orally once daily at the dose of 500mg of tepotinib hydrochloride hydrate.
  Arms: Tepotinib
Drug: Pemetrexed (Alimta) — 500 mg/m² every 3 weeks
  Arms: Investigator choice treatment
Drug: Vinorelbine — 25-30 mg/m² D1, D8, every 3 weeks
  Arms: Investigator choice treatment
Drug: Gemcitabine alone — 1250 mg/m² D1, D8, every 3 weeks
  Arms: Investigator choice treatment
Drug: Docetaxel — 75 mg/m² every 3 weeks
  Arms: Investigator choice treatment
Drug: Paclitaxel — 90 mg/m² D1, D8, D15 every 4 weeks If bevacizumab added: 10 mg/kg D1, D15 every 4 weeks
  Arms: Investigator choice treatment
Drug: Pembrolizumab — 200 mg every 3 weeks
  Arms: Investigator choice treatment
Drug: Nivolumab — 240 mg every 2 weeks
  Arms: Investigator choice treatment
Drug: Atezolizumab — 1200 mg every 3 weeks
  Arms: Investigator choice treatment

SUMMARY:
The hypothesize is that tepotinib is more effective than the investigator's choice of treatment in patients with MET-mutated NSCLC who have progressed after at least one first-line treatment.

The main benefit concerns patient access to tepotinib. There is currently no access to a new-generation MET TKI in France for METex14 patients, due to lack of comparative data. There are no phase III RCTs underway anywhere in the world. This study is the only opportunity, perhaps the last, to generate comparative data which, if positive, will enable the drug to be reimbursed. With this in mind, the methodology of this study was discussed with the HAS on several occasions beforehand, to ensure that it met their expectations. With a response rate of around 50% and a median progression-free survival of 11 months in previously-treated subjects based on clinical trials data, tepotinib is a key drug for METex14 NSCLC patients, who are generally elderly and frail, and for whom therapeutic options are limited.

The investigators expect to observe a benefit for patients treated with tepotinib compared to the control arm in terms of PFS, quality of life, objective response rate and duration of response. The overall survival benefit may be compromised by allowing patients in the control arm to cross over to tepotinib once they have progressed. However, the investigators have decided to maintain this crossover and consequently use PFS as the primary endpoint, as there is no clinical equipoise regarding the efficacy of tepotinib in METex14 NSCLC patients. The EMA has already approved tepotinib based on efficacy and safety data from clinical trials, and patients and investigators already consider this treatment as an important therapeutic option. Indeed, both ESMO and ASCO guidelines recommend the use of MET TKIs in these patients. In France, although neither tepotinib nor capmatinib are available, crizotinib, a multi-target TKI also active on MET, can be used off-label. If cross-over to tepotinib was not allowed in this trial, most patients would still benefit from cross-over to a MET TKI by receiving off-label crizotinib, which would in any case lead to a misinterpretation of the OS data. Therefore, the investigators believe it is preferable to control for cross-over and expose progressive patients in the control arm to tepotinib and use PFS as the primary endpoint.

Toxicity of MET TKIs is considered as manageable. In the VISION trial, of 313 patients treated with tepotinib (median age: 72 years), 109 (34.8%) experienced grade ≥3 treatment-related adverse events, leading to discontinuation in 46 patients (14.7%). Rates of adverse events (AE) were broadly consistent irrespective of prior therapies. Edema, the most common adverse event of clinical interest (AECI), was reported in 67.1% (grade ≥ 3, 11.2%). Median time to first edema onset was 7.9 weeks (range: 0.1-58.3). Edema was manageable with supportive measures, dose reduction (18.8%), and/or treatment interruption (23.1%), and rarely prompted discontinuation (4.3%). Other AECIs were also manageable and predominantly mild/moderate: hypoalbuminemia, 23.6% (grade ≥ 3, 3.5%); creatinine increase, 22.0% (grade ≥ 3, 1.0%); nausea, 23.3% (grade ≥ 3, 0.6%), diarrhea, 22.4% (grade ≥ 3, 0.3%), decreased appetite (grade ≥ 3, 0.3%), and ALT increase, 14.1% (grade ≥ 3, 2.2%). GI AEs typically occurred early and resolved in the first weeks10,13.

Given the efficacy of tepotinib, the manageable safety profile, and the oral administration of tepotinib, the investigators anticipate that treatment with tepotinib will be associated with improved quality of life.

Treatments offered in the control group correspond to standard treatments for advanced NSCLC in second line or beyond. In terms of prior lines of treatment, the eligibility criteria of the trial are aligned with the EMA label of tepotinib: "indicated for the treatment of adult patients with advanced non-small cell lung cancer (NSCLC) harboring alterations leading to MET gene exon 14 (METex14) skipping, who require systemic therapy following prior treatment with immunotherapy and/or platinum-based chemotherapy". The investigators have not included platinum-based chemotherapy as a treatment option in the control arm, considering that patients who are eligible to platinum-based chemotherapy should have received this regimen in first-line, as per ESMO guidelines14. Given the low efficacy of immunotherapy in patients with oncogene addiction, it is unlikely that some patients would receive immunotherapy alone as first-line treatment. Thus, the absence of platinum-based chemotherapy as a treatment choice in the control arm seems reasonable and will reduce the heterogeneity of this arm.

ELIGIBILITY:
Inclusion Criteria:

1. Informed, written and signed consent:

   * Patients must have signed and dated the written informed consent form approved by the ethics committee in accordance with the legal and institutional framework.
   * It must have been signed before protocol-related procedures that are not part of normal patient management are performed. Patients should be willing and able to adhere to the schedule of visits, treatment and laboratory tests.
2. Histologically proven advanced NSCLC.
3. Presence of a METex14 mutation (based on local testing). Detection of METex14 mutation should be performed on a tissue sample if available. In case no tissue sample is available, detection of METex14 on a liquid biopsy is authorized. The sponsor should be consulted if there is any doubt about the nature of the mutation.
4. Evidence of disease progression after at least one prior line of treatment including either a platinum-based chemotherapy or an anti-PD(L)1 agent or both.
5. Has received no more than 2 prior lines of treatment.
6. ECOG Performance Status 0-3.
7. Brain metastases are allowed. If immediate local treatment is required, inclusion is possible once the latter is complete.
8. Stage IIIB or IIIC non irradiable or stage IV (8th classification TNM, UICC 2015)
9. Age ≥ 18 years.
10. Adequate biological function:

    * Creatinine clearance ≥ 30 ml/min;
    * Neutrophils ≥ 1500/mm3;
    * Platelets ≥100,000/mm3;
    * Haemoglobin ≥ 8 g/dL;
    * Liver enzymes < 3x ULN except for patients with liver metastases (< 5x ULN);
    * Total bilirubin ≤ 1.5 x ULN except for patients with proven Gilbert's syndrome (≤ 5 x ULN) or patients with liver metastases (≤ 3.0 ULN).
11. Protected adults may participate in the study if they are capable of making decisions regarding their medical treatment in accordance with the guardianship judgment.
12. For women of childbearing potential (including women who have had a tubal ligation), serum pregnancy test must be performed and documented as negative within 14 days prior to C1D1.
13. Women of childbearing potential must remain abstinent (refrain from heterosexual intercourse) or use contraceptive methods with a failure rate of < 1% per year during the treatment period and for at least 6 months after the last dose of study drugs. Women must refrain from donating eggs during this same period. A woman is considered to be of childbearing potential if she is post-menarcheal, has not reached a postmenopausal state (≥ 12 continuous months of amenorrhea with no identified cause other than menopause), and has not undergone surgical sterilization (removal of ovaries or uterus). Examples of contraceptive methods with a failure rate of <1% per year include bilateral tubal ligation, male sterilization, established proper use of hormonal contraceptives that inhibit ovulation, hormone-releasing intrauterine devices, and copper intrauterine devices. Hormonal contraceptive methods must be supplemented by a barrier method plus spermicide. The reliability of sexual abstinence should be evaluated in relation to the duration of the clinical study and the preferred and usual lifestyle of the patient. Periodic abstinence (e.g. calendar, ovulation, symptothermal, or postovulation methods) and withdrawal are not acceptable methods of contraception.
14. Men with female partners of childbearing potential or pregnant female partners, must remain abstinent or use a condom during the treatment period and for at least 6 months after the last dose of study treatment to avoid exposing the embryo. Men must refrain from donating sperm during this same period. The reliability of sexual abstinence should be evaluated in relation to the duration of the clinical study and the preferred and usual lifestyle of the patient. Periodic abstinence (e.g. calendar, ovulation, symptothermal, or postovulation methods) and withdrawal are not acceptable methods of contraception.
15. Patient covered by a national health insurance.

Exclusion Criteria:

1. Prior treatment with a MET inhibitor (including crizotinib).
2. Presence of another known driver oncogene alteration (including EGFR, HER2, KRAS, BRAF mutations or ALK, ROS1, RET fusions). In case of detection of any other driver alteration, inclusion should be discussed with the sponsor.
3. ECOG Performance Status 4.
4. Known hypersensitivity to tepotinib or its excipients.
5. History of cancer within 3 years or active cancer except those with a negligible risk of metastasis or death, or those treated curatively. If a patient does not fulfil this criterion but the investigator considers that the benefit/risk balance is in favour of inclusion in the study, please contact IFCT.
6. Inability to comply with study or follow-up procedures.
7. Pregnant, lactating, or breastfeeding women.
8. Any disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug, that may affect the interpretation of the results, or that may render the patient at high risk from treatment complications.
9. History of idiopathic pulmonary fibrosis or active pneumonitis on chest computed tomography (CT) scan at screening. History of radiation pneumonitis in the radiation field (fibrosis) is permitted.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 133 (Estimated)
Dates: Start 2025-12-09 (Actual); Primary Completion 2028-03-15 (Estimated); Study Completion 2028-07-15 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) | About 36 months
  Progression-free survival is calculated from the date of randomization until progression as defined by independent review comity according to RECIST 1.1 or death (whichever occurs first).

SECONDARY OUTCOMES:
Global Health Status Quality of life | 6 weeks after randomization
  Quality of life will be assessed using the EORTC (European Organisation for Research and Treatment of Cancer) Quality of Life Questionnaire C30 with lung cancer module LC29 at baseline and week 6. A linear transformation will be applied to standardise the raw score to a 0-100 range (100=best possible QoL). A 10-point change will be considered clinically meaningful.
Overall Survival | About 36 months
  Overall survival is calculated from the date of randomization until death (for whatever reason).
Second Progression-Free Survival (PFS2) | About 36 months
  PFS2 is defined as the time from randomization to the date of progression of disease on first subsequent systemic anti-cancer therapy (as defined by the RECIST criteria v.1.1) (second progression), or death from any cause, whichever occurs first.
Time to next treatment or death (TNT-D) | About 36 months
  TNT-D is defined as the time from randomization to the date of first subsequent systemic anti-cancer therapy (as defined by the RECIST criteria v.1.1), or death from any cause, whichever occurs first.
Objective Response Rate (ORR) | About 36 months
  ORR is defined as the proportion of patients who have achieved a best overall response of complete response (CR) or partial response (PR) as determined by investigator review of radiographic disease assessments per RECIST v1.1.
Duration of response (DOR) | About 36 months
  DOR is defined as the time from the date of the first documented response (CR or PR) to the earliest date of disease progression, as determined by Investigator review of radiographic disease assessments per RECIST v1.1, or death due to any cause.
Quality of life of patient | About 36 months
  Quality of life will be assessed using the EORTC (European Organisation for Research and Treatment of Cancer) C30 with lung cancer module LC29 at baseline and week 6. For each scale in QLQ-C30 LC29, a linear transformation will be applied to standardise the raw score to a 0-100 range (100=best possible function or QoL for functional scales and highest symptom burden for symptom scales and symptom items). A 10-point change in an item or domain will be considered clinically meaningful. QoL will be defined as improved when a ≥10-point increase will be recorded for functioning scales and ≥10-point reduction for symptom domains.
Observance of treatments | About 36 months
  The number of cycles will be reported for each arm. The number of dose interruptions and dose modifications will be reported on the safety population.
Safety and tolerability of treatments | About 36 months
  Safety is measured by the frequency and the severity of adverse events, serious or not, at each patient visit and at each post treatment follow-up visit using the CTCAE Version 5.0.

CONTACTS AND LOCATIONS:
Locations (29):
- France (29):
  - Besançon - CHU, Besançon
  - Bordeaux - Institut Bergonie, Bordeaux
  - Brest - CHU, Brest
  - Caen - CRLCC, Caen
  - Centre Hospitalier Intercommunal de Créteil, Créteil
  - Dijon - Centre Georges-François Leclerc, Dijon
  - Grenoble - CHU, Grenoble
  - CHD Vendée, La Roche-sur-Yon
  - Le Mans - CHG, Le Mans
  - CHRU de Lille, Lille
  - Centre Léon Bérard, Lyon
  - Institut Paoli Calmette, Marseille
  - Marseille - APHM, Marseille
  - Montpellier - CHU, Montpellier
  - Centre Antoine Lacassagne, Nice
  - AP-HP Hôpital Cochin, Paris
  - AP-HP Hôpital Tenon, Paris
  - Paris - APHP Bichat, Paris
  - Centre Hospitalier Général - Pau, Pau
  - Bordeaux - CHU, Pessac
  - Institut de Cancérologie de l'Ouest - René Gauducheau, Saint-Herblain
  - Sens - CH, Sens
  - Strasbourg - NHC, Strasbourg
  - Toulon - CHI, Toulon
  - CHU Toulouse, Toulouse
  - CHRU de Tours, Tours
  - CH de Valence, Valence
  - Nancy - CHU, Vandœuvre-lès-Nancy
  - Gustave Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: Yes
The individual participant data underlying the results reported in this article, as well as the study protocol and statistical analysis plan, will be made available after deidentification immediately following publication and for three years. Researchers who provide a methodologically sound proposal for any purpose may direct proposals to contact@ifct.fr. To gain access, data requestors will need to sign a data access agreement that requires approval by the French Cooperative Thoracic Intergroup.

REFERENCES:
- See also: IFCT website — https://www.ifct.fr/etudes-cliniques/1239-ifct-etude2404